CLINICAL TRIAL: NCT03053128
Title: Implication of Cardiac Shock Wave Therapy on Coronary Artery Disease: A Prospective Randomized Double-blind Control Trial
Brief Title: Implication of Cardiac Shock Wave Therapy on Coronary Artery Disease
Acronym: CSWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Qing He, Cinical professor and Principal investigator, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-2016004
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Ischemia
Keywords: cardiac ischemia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSWT group (Experimental): Patients in CSWT group will receive cardiac shock wave therapy for three moths, every first week of the month.
  Interventions: Device: Cardiac shock wave therapy
- Sham CSWT group (Sham Comparator): Patients in sham CSWT group will receive sham cardiac shock wave, which segregated by an air-cushion.
  Interventions: Other: Sham cardiac shock wave (Control group)

INTERVENTIONS:
Device: Cardiac shock wave therapy — Patients in CSWT group will receive CSWT for a 3-month therapy, located in their ischemia area with a energy of 0.09mJ/mm2. Patients will get therapy on every first week of the month and rest for following three weeks.
  Other Names: CSWT group
  Arms: CSWT group
Other: Sham cardiac shock wave (Control group) — Patients in sham CSWT group will receive sham cardiac shock wave, which is segregated by an air cushion.
  Other Names: Sham CSWT group
  Arms: Sham CSWT group

SUMMARY:
Coronary heart disease (CHD) is a public health care challenge. There are three types of treatment for CHD, medication, percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG). However, some end-stage CHD patients lost the chance to get those treatment. Cardiac shock wave therapy (CSWT) is a new developed therapy for these patients, which is used in tens of countries all over the world. Safety, invasiveness, effectiveness is its advantage. Ischemia condition can be improved after CSWT. There are only three cities in China run the program of CSWT, which are Kunming, Beijing and Shanghai. The investigators designed a randomized double-blind study to evaluate the effectiveness and safety of CSWT.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is a public health care challenge, which lead to 3.5 millions of people died in China every year. There are three types of treatment for CHD, medication, percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG). However, some end-stage CHD patients with severe cardiac ischemia lost the chance to get those treatment. Their quality of life is influenced by recurrent angina. Cardiac shock wave therapy (CSWT) is a new developed therapy for these patients, which is used in tens of countries all over the world. German and Japan are the countries earliest used CSWT. Safety, invasiveness, effectiveness is its advantage. Ischemia condition can be improved after CSWT by objective examination. New small vessels generation on ischemia area was found on mice and pig model. There are only three cities in China run the program of CSWT, that are Kunming, Beijing and Shanghai. Beijing hospital has the only CSWT machine in Beijing. The investigators designed a randomized double-blind study to evaluate the effectiveness and safety of CSWT.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple or diffused coronary artery stenosis by coronary angiography and not candidate for PCI or CABG;
2. Myocardial ischemia and/or cardiac dysfunction by objective exams;
3. Angina and/or heart failure could not be control after optimal medication treatment for coronary artery disease;
4. LVEF is above 30%;
5. Signed informed consent

Exclusion Criteria:

1. Acute myocardial infarction;
2. Within one month after PCI or CABG;
3. Heart transplant patient;
4. Mechanic valve implantation patient;
5. Uncontrolled heart failure with LVEF less than 30%;
6. Severe arrhythmia;
7. Pacemaker implantation patient;
8. Infective endocarditis;
9. Severe chronic obstructive pulmonary disease patient;
10. Pregnant or nursing patient;
11. Silicone breast forms patient;
12. Chest tumor patient;
13. Participant in other clinical trials at the same time.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion score | 1st week of fourth month from beginning of CSWT
  Myocardial perfusion score will be calculated by myocardial perfusion imaging though single-photon computer tomography.
Ischemia area percentage | 1st week of fourth month from beginning of CSWT
  Ischemia area will be calculated by myocardial perfusion imaging though single-photon computer tomography.

SECONDARY OUTCOMES:
Cardiac wall motion amplitude | 1st week of fourth month from beginning of CSWT
  Cardiac wall motion amplitude rate will be calculated by single-photon computer tomography.
Left ventricular thickness rate | 1st week of fourth month from beginning of CSWT
  Left ventricular thickness rate will be calculated by single-photon computer tomography.
Cardiac enzyme | First week after CSWT
  Troponin T and troponin I will be tested at last time shock wave therapy of the first week.
Angina score-SAQ | 1st week of fourth month from beginning of CSWT
  SAQ angina score will be finished after three month of CSWT.
Quality of life (SF-36) | 1st week of fourth month from beginning of CSWT
  SF-36 questionnaire will be used for QOL.
Six-minute of walk test | 1st week of fourth month from beginning of CSWT
  6MWT will be used for exertional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Qing He, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu W, Shen T, Liu B, Wang S, Li J, Dai D, Cai J, He Q. Cardiac shock wave therapy attenuates H9c2 myoblast apoptosis by activating the AKT signal pathway. Cell Physiol Biochem. 2014;33(5):1293-303. doi: 10.1159/000358697. Epub 2014 Apr 28. PMID 24802592